CLINICAL TRIAL: NCT01838668
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of BG00012 in Subjects From the Asia-Pacific Region and Other Countries With Relapsing-Remitting Multiple Sclerosis
Brief Title: An Efficacy and Safety Study of BG00012 (Dimethyl Fumarate) in Asian Subjects With Relapsing Remitting Multiple Sclerosis (RRMS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109MS305; 2013-004533-32 (EudraCT Number)
Record Dates: First submitted 2013-04-20; First posted 2013-04-24 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part I Placebo (Placebo Comparator): Placebo orally twice a day. In Part I: participants will be randomized into one of 2 groups: BG00012, 240 mg twice daily (BID) or matching placebo BID
  Participants will begin the study by taking 1 capsule orally BID for first 7 days and escalate their dosing from day 8 to 2 matching capsules orally BID.
  Interventions: Drug: Placebo
- Part I BG00012 (Experimental): BG00012 240 mg orally twice a day (participants will begin dosing at 120 mg BG00012 twice daily (BID) for the first 7 days and 240 mg BG00012 BID thereafter.) In Part I: participants will be randomized into one of 2 groups: BG00012, 240 mg twice daily (BID) or matching placebo BID
  Interventions: Drug: dimethyl fumarate
- Part II BG00012 (Experimental): Part II: All participants will receive BG00012 240 mg orally twice a day (participants will begin dosing at 120 mg (1 capsule) BG00012 twice daily (BID) for the first 7 days and 240 mg (2 capsules) BG00012 BID thereafter.
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: Placebo — Two placebo capsules orally BID
  Arms: Part I Placebo
Drug: dimethyl fumarate — Two dimethyl fumarate 120mg capsules orally BID
  Other Names: BG00012; Tecfidera; DMF
  Arms: Part I BG00012; Part II BG00012

SUMMARY:
This is a multicenter study conducted in 2 parts:

The primary objective in Part I of this study is to determine the efficacy of BG00012 (dimethyl fumarate, DMF) on inflammatory brain magnetic resonance imaging (MRI) lesion activity (Gadolinium-enhancing lesions) when compared with placebo from 4 scans performed at Weeks 12, 16, 20, and 24 in participants with Relapsing Remitting Multiple Sclerosis (RRMS) including participants from the Asia-Pacific region.

The secondary objectives in Part I of this study in this study population are to determine whether BG00012, when compared with placebo over 24 weeks, is effective in reducing the cumulative number of new Gadolinium-enhancing lesions from Baseline to Week 24; reducing the number of new or newly enlarging T2 hyperintense lesions on brain MRI scans at Week 24 compared with Baseline.

The primary objective in Part II (open label) of this study is to evaluate the long-term safety profile of BG00012 in eligible participants from Part I.

ELIGIBILITY:
Key Inclusion Criteria:

* Inclusion Criteria for Part I:

  * Must have a diagnosis of Relapsing-Remitting Multiple Sclerosis (RRMS).
  * Must have a baseline Expanded Disability Status Scale (EDSS) score between 0.0 and 5.0, inclusive.

Key Inclusion Criteria for Part II:

• Subjects who participated in and completed Part I per protocol.

Key Exclusion Criteria:

* Other chronic disease of the immune system, malignancies, acute urologic, pulmonary, gastrointestinal disease.
* Pregnant or nursing women.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2015-06-16 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Total number of new Gadolinium-enhancing lesions over 4 scans at Weeks 12, 16, 20, and 24. | Part I (Week 24)
Incidence of treatment-emergent adverse events and serious adverse events | Part II (Up to 4.5 years)

SECONDARY OUTCOMES:
Cumulative number of new Gadolinium-enhancing lesions from Baseline to Week 24 | Part I (Week 24)
Number of new or newly enlarging T2 hyperintense lesions at Week 24 compared with Baseline | Part I (Week 24)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (54):
- Czechia (9):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Neurospol, s.r.o., Havířov
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Privatni ordinace - neurologie, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni poliklinika VFN, Prague
  - Fakultni nemocnice v Motole, Prague
  - Krajska zdravotni, a.s. - Nemocnice Teplice, o.z., Teplice
- Japan (27):
  - NHO Asahikawa Medical Center, Asahikawa-shi
  - Juntendo University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Kanazawa Medical University Hospital, Kahoku-gun
  - Saitama Medical Center, Kawagoe-shi
  - Kobe University Hospital, Kobe
  - National Center Hospital, NCNP, Kodaira-shi
  - Kyoto University Hospital, Kyoto
  - NHO Utano Hospital, Kyoto
  - Iwate Medical University Hospital, Morioka
  - Niigata University Medical & Dental Hospital, Niigata
  - Irino Clinic, Inc., Osaka
  - Kindai University Hospital, Osakasayama-shi
  - Tokyotohokeniryokosya Ebara Hospital, Ōta-ku
  - NHO Hokkaido Medical Center, Sapporo
  - CEReS Sapporo Neurology Clinic, Sapporo
  - Tohoku University Hospital, Sendai
  - Keio University Hospital, Shinjuku-ku
  - Department of Neurosurgery, Tokyo Women's Medical University, Shinjuku-ku
  - Osaka University Hospital, Suita-shi
  - National Defense Medical College Hospital, Tokorozawa-shi
  - Ehime University Hospital, Toon-shi
  - Tsukuba University Hospital, Tsukuba
  - Yamaguchi University Hospital, Ube-shi
  - Tokyo Womens Medical University Yachiyo Medical Center, Yachiyo-shi
  - Yokohama City University Hospital, Yokohama
- Poland (9):
  - Copernicus Podmiot Leczniczy Sp. z o.o., Gdansk
  - M.A. - LEK A.M.Maciejowscy SC., Katowice
  - Nzoz Novo-Med, Katowice
  - Neuro-Care Gabriela Klodowska, Katowice
  - MCD Medical, Krakow
  - Centrum Neurologii K. Selmaj, Lodz
  - Neurologiczny NZOZ Centrum Leczenia SM, Plewiska
  - NZOZ "NEURO-KARD", "Ilkowski i Partnerzy" Sp. Partn. Lek., Poznan
  - Miedzyleski Szpital Specjalistyczny, Warsaw
- South Korea (6):
  - Yeungnam University Hospital, Daegu
  - National Cancer Center, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Kondo T, Kawachi I, Onizuka Y, Hiramatsu K, Hase M, Yun J, Matta A, Torii S. Efficacy of dimethyl fumarate in Japanese multiple sclerosis patients: interim analysis of randomized, double-blind APEX study and its open-label extension. Mult Scler J Exp Transl Clin. 2019 Jul 31;5(3):2055217319864974. doi: 10.1177/2055217319864974. eCollection 2019 Jul-Sep. PMID 31391949
- [Derived] Saida T, Yamamura T, Kondo T, Yun J, Yang M, Li J, Mahadavan L, Zhu B, Sheikh SI. A randomized placebo-controlled trial of delayed-release dimethyl fumarate in patients with relapsing-remitting multiple sclerosis from East Asia and other countries. BMC Neurol. 2019 Jan 7;19(1):5. doi: 10.1186/s12883-018-1220-3. PMID 30616596
- [Derived] Ochi H, Niino M, Onizuka Y, Hiramatsu K, Hase M, Yun J, Matta A, Torii S. 72-Week Safety and Tolerability of Dimethyl Fumarate in Japanese Patients with Relapsing-remitting Multiple Sclerosis: Analysis of the Randomised, Double Blind, Placebo-Controlled, Phase III APEX Study and its Open-Label Extension. Adv Ther. 2018 Oct;35(10):1598-1611. doi: 10.1007/s12325-018-0788-8. Epub 2018 Sep 11. PMID 30206820
- See also: EudraCT Tabulated Result — https://www.clinicaltrialsregister.eu/ctr-search/trial/2013-004533-32/results